CLINICAL TRIAL: NCT03342963
Title: A Single-center, Open-label, Randomized, Two-treatment, Two-period Crossover Trial to Investigate Bioequivalence Between Single Administration of ASC-01 (Aripiprazole/Sertraline Combination Drug) and Concomitant Single Administration of Aripiprazole and Sertraline, and Food Effect on Pharmacokinetics of ASC-01 in Healthy Male Adults
Brief Title: Bioequivalence Between Single Administration of ASC-01 (Aripiprazole/Sertraline Combination Drug) and Concomitant Single Administration of Aripiprazole and Sertraline, and Food Effect on Pharmacokinetics of ASC-01 in Healthy Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 031-102-00214; JapicCTI-173774 (Other: Japic)
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Healthy Male Adults
MeSH Terms: interventions — Aripiprazole; Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASC-01 in period 1, Aripiprazole and sertraline in period 2 (Experimental): At Day 1 in Period I, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) will be administered after 10 or more hours of fasting.
  At Day 1 in Period II, Aripiprazole 3 mg and sertraline 100 mg will be administered after 10 or more hours of fasting.
  Interventions: Drug: ASC-01; Drug: Aripiprazole and sertraline
- Aripiprazole and sertraline in period 1, ASC-01 in period 2 (Experimental): At Day 1 in Period I, Aripiprazole 3 mg and sertraline 100 mg will be administered after 10 or more hours of fasting.
  At Day 1 in Period II, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) will be administered after 10 or more hours of fasting.
  Interventions: Drug: ASC-01; Drug: Aripiprazole and sertraline
- Fasting in period 1, After breakfast in period 2 (Experimental): At Day 1 in Period I, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) will be administered after 10 or more hours of fasting.
  At Day 1 in Period II, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) will be administered 30 minutes after the start of breakfast.
  Interventions: Drug: ASC-01; Drug: Aripiprazole and sertraline
- After breakfast in period 1, Fasting in period 2 (Experimental): At Day 1 in Period I, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) will be administered 30 minutes after the start of breakfast.
  At Day 1 in Period II, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) will be administered after 10 or more hours of fasting.
  Interventions: Drug: ASC-01; Drug: Aripiprazole and sertraline

INTERVENTIONS:
Drug: ASC-01 — Aripiprazole 3 mg/sertraline 100 mg combination drug
Drug: Aripiprazole and sertraline — Aripiprazole 3 mg and sertraline 100 mg

SUMMARY:
To investigate the bioequivalence of aripiprazole between administration of one ASC-01 tablet (aripiprazole 3 mg/sertraline 100 mg combination drug) and concomitant administration of one aripiprazole 3-mg tablet and two sertraline 50-mg tablets (Cohort 1).

To investigate food effect on plasma pharmacokinetics of aripiprazole and sertraline by single oral administration of ASC-01 under a fasting or fed condition (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject at the age between 20 and 40 at the time of informed consent
* Subject has a body mass index (BMI = body weight [kg]/height [m]2) of ≥18.5 and <25.0 kg/m2 at screening
* Subject is providing consent for participation in this trial in writing prior to the start of the procedures related to this trial, and judged by the investigator or subinvestigator to be capable of observing procedures in this trial.

Exclusion Criteria:

* Subject has a clinically significant abnormality in physical findings at screening or in medical history that in the investigator's or subinvestigator's opinion may place the subject at risk or interfere with outcome variables including drug absorption, distribution, metabolism, and excretion.
* Subject is judged by the investigator or subinvestigator to be inappropriate for participation in this trial.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of Kyusyu Region, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: ASC-01 First: At Day 1 in Period I, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) was administered after 10 or more hours of fasting.
  At Day 1 in Period II, Aripiprazole 3 mg and sertraline 100 mg was administered after 10 or more hours of fasting.
  There was a washout period of at least 35 days between Period I and Period II.
- Cohort 1: Aripiprazole/Sertraline Concomitant First: At Day 1 in Period I, Aripiprazole 3 mg and sertraline 100 mg was administered after 10 or more hours of fasting.
  At Day 1 in Period II, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) was administered after 10 or more hours of fasting.
  There was a washout period of at least 35 days between Period I and Period II.
- Cohort 2: ASC-01 Under Fasted First: At Day 1 in Period I, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) was administered after 10 or more hours of fasting.
  At Day 1 in Period II, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) was administered 30 minutes after the start of breakfast.
  There was a washout period of at least 35 days between Period I and Period II.
- Cohort 2: ASC-01 Under Fed First: At Day 1 in Period I, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) was administered 30 minutes after the start of breakfast.
  At Day 1 in Period II, ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) was administered after 10 or more hours of fasting.
  There was a washout period of at least 35 days between Period I and Period II.
Period: Overall Study
Arm/Group | Cohort 1: ASC-01 First | Cohort 1: Aripiprazole/Sertraline Concomitant First | Cohort 2: ASC-01 Under Fasted First | Cohort 2: ASC-01 Under Fed First
Started | 27 | 27 | 10 | 10
Completed | 25 | 25 | 10 | 10
Not Completed | 2 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set: subjects who received investigational medicinal product (IMP) at least once.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ASC-01 First | Cohort 1: Aripiprazole/Sertraline Concomitant First | Cohort 2: ASC-01 Under Fasted First | Cohort 2: ASC-01 Under Fed First | Total
Number analyzed (Participants) | 27 | 27 | 10 | 10 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 10 | 10 | 74
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 27 | 27 | 10 | 10 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 27 | 27 | 10 | 10 | 74
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 27 | 27 | 10 | 10 | 74

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax) of Aripiprazole in Cohort 1
Time Frame: Baseline, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72,96, 144 and 168h after dosing
Population: Pharmacokinetic Analysis Set comprised subjects who received IMP and for whom plasma drug concentration data were obtained.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ASC-01: ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) was administered after 10 or more hours of fasting.
- Aripiprazole/Sertraline Concomitant: Aripiprazole 3 mg and sertraline 100 mg was administered after 10 or more hours of fasting.
Arm/Group | ASC-01 | Aripiprazole/Sertraline Concomitant
Number analyzed (Participants) | 40 | 39
ng/mL | 18.8 (5.33) | 16.9 (4.38)

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve 168h (AUC168h) of Aripiprazole in Cohort 1
Time Frame: Baseline, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72,96, 144 and 168h after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ASC-01 | Aripiprazole/Sertraline Concomitant
Number analyzed (Participants) | 40 | 39
ng*h/mL | 783 (273) | 779 (236)

3. Primary Outcome: Cmax of Aripiprazole and Sertraline in Cohort 2
Time Frame: Baseline, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72,96, 144 and 168h after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ASC-01 Under Fasted: ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) was administered after 10 or more hours of fasting.
- ASC-01 Under Fed: ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) was administered 30 minutes after the start of breakfast.
Arm/Group | ASC-01 Under Fasted | ASC-01 Under Fed
Number analyzed (Participants) | 20 | 20
ng/mL
  Aripiprazole: number analyzed (Participants) | 16 | 11
  Aripiprazole | 16.9 (5.23) | 16.6 (3.74)
  Sertraline: number analyzed (Participants) | 14 | 11
  Sertraline | 28.9 (10.7) | 36.5 (15.6)

4. Primary Outcome: AUC168h of Aripiprazole and Sertraline in Cohort 2
Time Frame: Baseline, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72,96, 144 and 168h after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ASC-01 Under Fasted | ASC-01 Under Fed
Number analyzed (Participants) | 20 | 20
ng*h/mL
  Aripiprazole: number analyzed (Participants) | 16 | 11
  Aripiprazole | 701 (221) | 865 (219)
  Sertraline: number analyzed (Participants) | 14 | 11
  Sertraline | 904 (415) | 1060 (468)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events occurring up to 8 days after dosing date were collected.
Description: Safety Set comprised subjects who received IMP at least once.
Groups:
- Cohort 1 - ASC-01; Cohort 2 - ASC-01 Under Fasted: ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) was administered after 10 or more hours of fasting.
- Cohort 1 - Aripiprazole/Sertraline Concomitant: Aripiprazole 3 mg and sertraline 100 mg was administered after 10 or more hours of fasting.
- Cohort 2 - ASC-01 Under Fed: ASC-01 (aripiprazole 3 mg/sertraline 100 mg combination drug) was administered 30 minutes after the start of breakfast.
Arm/Group | Cohort 1 - ASC-01 | Cohort 1 - Aripiprazole/Sertraline Concomitant | Cohort 2 - ASC-01 Under Fasted | Cohort 2 - ASC-01 Under Fed
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 44/52 | 43/52 | 12/20 | 14/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - ASC-01 (N=52) | Cohort 1 - Aripiprazole/Sertraline Concomitant (N=52) | Cohort 2 - ASC-01 Under Fasted (N=20) | Cohort 2 - ASC-01 Under Fed (N=20)
Tachycardia (Cardiac disorders) | 3 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 9 | 3 | 1
Nausea (Gastrointestinal disorders) | 39 | 38 | 11 | 10
Vomiting (Gastrointestinal disorders) | 20 | 17 | 6 | 9
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT03342963/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT03342963/SAP_001.pdf